CLINICAL TRIAL: NCT04315597
Title: Doubleblind, Randomized, Placebo-controlled, Multicenter Clinical Study to Investigate Relaps-prevention by Hypericumextract in Outpatients With Moderate Depressive Episodes (Major Depression)
Brief Title: Study to Learn About Relapse Prevention of Hypericumextract (a Drug Based on the Plant St. John Wort) in Outpatients Suffering From Moderate Depressive Episodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Steigerwald Arzneimittelwerk GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20997; 2008-001417-26 (EudraCT Number)
Record Dates: First submitted 2020-03-05; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Moderate Depressive Episodes (Major Depression)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypericum extract STW 3-VI (Laif® 900, BAY98-7108) (Experimental)
  Interventions: Drug: Laif® 900, BAY98-7108
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Laif® 900, BAY98-7108 — 1 x daily, 1 tablet, 900 mg
  Arms: Hypericum extract STW 3-VI (Laif® 900, BAY98-7108)
Drug: Placebo — 1 x daily, 1 tablet, 900 mg
  Arms: Placebo

SUMMARY:
The researchers in this trial want to learn more about the drug Laif® 900 in preventing the return of signs and symptoms of depressions (also called relapse) in patients suffering from moderate depression episodes. The study drug Laif® 900 is based on Hypericumextract made from the plant St. John wort. Patients will be accepted to take part in the study if they have 20-24 points on the Hamilton Depression Rating Scale (HAM-D) which is a questionnaire helping the doctor to rate the severity of the depression and includes questions on patient's mood, sleep difficulties, agitation, anxiety and weight loss. About 400 patients will be enrolled into the first part of the study and will be treated for 12 weeks with Laif® 900 capsule once daily. Only patients with an improved HAM-D score by 50% will stay in the study and continue with the second part of the study which will last for 24 weeks.

In this second part of the study patients will receive either Laif® 900 capsule once daily or an inactive tablet (placebo). Neither the treating doctor nor the patient will know which patient receives the Laif® 900 or placebo. At the end of the study the researcher will assess the effectiveness of the study drug in prevention relapse of depression episodes and will also have more information on the safety of the study drug.

ELIGIBILITY:
Inclusion Criteria:

Study Phase 1:

* Age 18-70 years
* Diagnosis according to DSM-IV-TR: 296.32: Outpatients with a mediocre depressive episode requiring treatment for recurrent major depression
* At least 5 of the following symptoms must persist for 2 weeks, with at least one of the main symptoms:
* Depressed mood (main symptom)
* Loss of interest or pleasure (main symptom)
* Significant weight loss without diet or weight gain
* Increased sleep or insomnia
* Psychomotor restlessness or slowing down
* Excessive, inappropriate guilt or feelings of worthlessness on almost every day
* Subjective or observable diminished ability to think and to decide
* Fatigue and loss of energy
* Suicidal thoughts and / or actions

Study Phase 2:

* Phase 1 responders (= Phase 1 patients who have at least a 50% decrease in the HAMD-17 total score after 12 weeks of Laif® 900 therapy).

Exclusion Criteria: General (phase 1 and phase 2)

* Unable to work and patients cared for according to the BtG (working group "Stay") and "Medical Measures")
* Simple mourning reaction
* Clinically relevant laboratory abnormalities due to severe organ and systemic diseases
* Taking immunosuppressants (eg after organ transplants)
* Taking oral contraceptives with low levels of hormones (estrogen ≤ 50 μg, micropillus)
* Thyroid dysfunction (patients with non-euthyroid TSH levels)
* Known intolerance to the test medication
* Known photosensitivity
* Diabetes mellitus type I and II requiring treatment
* Unstable hypertension
* Pregnancy or breastfeeding
* Cancer and AIDS patients (HIV-positive)
* Alcohol, drug or drug abuse in the last 6 months
* Coadministration with coumarin-type anticoagulants
* History of epilepsy
* Melanoma
* Specific psychotherapy in the last 2 months and during the clinical trial
* Participation in a clinical trial within the last 30 days
* Simultaneous participation in another clinical trial
* Compliance and protocol management are not guaranteed by language problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2009-03-03 (Actual); Primary Completion 2011-11-22 (Actual); Study Completion 2011-11-22 (Actual)

PRIMARY OUTCOMES:
Relapse rate | 24 weeks
  Definition: Increase of the Hamilton rating scale for depression (HAMD)-17 total score in Phase 2 by > 5 points compared to Phase 2 baseline, if at the same time a total score of at least 12 is reached.

SECONDARY OUTCOMES:
Time between baseline and occurrence of relaps measured by: Total score of HAMD-17 | 24 weeks
Time between baseline and occurrence of relaps measured by: Beck Depression Inventory (BDI) | 24 weeks
Time between baseline and occurrence of relaps measured by: Clinical Global Impressions (CGI) | 24 weeks
Global assessment of efficacy by investigators and patients | 12 and 24 weeks
  % of investigators and patients, respectively, who rated the efficacy "very good" or "good", respectively.
Safety and Tolerability: Number of Adverse Events | 36 weeks

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.